CLINICAL TRIAL: NCT03172130
Title: Prospective Study of Efficacy of Sham CPAP vs. Straight CPAP on Cough Intensity in Patients With Chronic Cough
Brief Title: Sham CPAP vs. Straight CPAP for Chronic Cough
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Krishna M. Sundar (Other)
Responsible Party: Sponsor-Investigator, Krishna M. Sundar, Principal Investigator, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB #62049
Record Dates: First submitted 2017-05-27; First posted 2017-06-01 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-06

CONDITIONS: Chronic Cough; OSA
Keywords: Obstructive Sleep Apnea; CPAP
MeSH Terms: conditions — Chronic Cough; Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Straight CPAP (Experimental): Patients randomized to straight CPAP will receive 10 cm of air pressure, or as determined by the results of polysomnography, for 6 weeks. Following the 6-week visit, patients will be placed on straight CPAP with equipment approved by insurance for an additional 6 weeks.
  Interventions: Device: Straight CPAP
- Sham CPAP (Sham Comparator): Patients randomized to sham CPAP will receive 1-2 cm of air pressure for 6 weeks. Following the 6-week visit, patients will be placed on straight CPAP with equipment approved by insurance for an additional 6 weeks.
  Interventions: Device: Sham CPAP

INTERVENTIONS:
Device: Straight CPAP
  Arms: Straight CPAP
Device: Sham CPAP
  Arms: Sham CPAP

SUMMARY:
Chronic cough is an important clinical problem in primary care and sub-specialty practice. Besides the distress experienced by patients with chronic cough, significant healthcare resources are expended to understand the role of gastroesophageal reflux, asthma and post-nasal drip in understanding their contribution to cough.

Obstructive sleep apnea (OSA) is common in patients with chronic cough. More importantly, treatment of OSA with continuous positive airway pressure (CPAP) has led to improvement in cough for chronic cough patients. Mechanisms by which OSA therapy with CPAP can improve cough includes beneficial effects on reflux and airway inflammation.

The aim of this study is to definitively establish that CPAP therapy for treatment of OSA in chronic cough patients improves cough. While these patients with chronic cough are not routinely screened and treated for OSA, this study aims to evaluate these chronic cough patients with screening questionnaires for OSA and if necessary with polysomnography and randomize them to either CPAP or sham CPAP for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Cough of more than 2 month duration
* Not active smoker with history of stoppage of smoking for more than 6 months
* Evaluation and treatment by other providers for suspected gastroesophageal reflux disease (GERD), upper airway cough syndrome (UACS), or cough-variant asthma (CVA) for at least 1 month
* Normal chest radiography or computed tomography (CT) scans (patients with up to 2 lung nodules less than 3 mm will be allowed if there is no history of malignancy elsewhere)
* Normal spirometry with predicted diffusing capacity of the lung for carbon dioxide (DLCO) more than 50% predicted. Pulmonary Function Test criteria: no evidence of airflow limitation (FEV1/FVC > 0.7) or significant chest restriction (FVC > 70% predicted) with predicted DLCO more than 50% predicted

Exclusion Criteria:

* Pregnancy
* Recent pneumonia (less than 6 months)
* Congestive heart failure, acute or chronic renal disease, jaundice or chronic liver disease, pulmonary embolism, stroke or neurodegenerative disease, malignancy
* Use of supplemental oxygen or positive airway pressure therapy (if patients have been diagnosed with obstructive sleep apnea in the past but were non-compliant with positive airway pressure therapy, they will not be excluded)
* Use of opiates for cough suppression (opiate use for pain suppression can be included)
* Alcoholism, drug dependence (including chewing tobacco) or illicit drug use
* Esophageal cancer or laryngeal surgery
* Craniofacial abnormalities that preclude CPAP placement

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-10-13 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krishna Sundar, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sundar KM, Willis AM, Smith S, Hu N, Kitt JP, Birring SS. A Randomized, Controlled, Pilot Study of CPAP for Patients with Chronic Cough and Obstructive Sleep Apnea. Lung. 2020 Jun;198(3):449-457. doi: 10.1007/s00408-020-00354-1. Epub 2020 Apr 30. PMID 32356074

RESULTS

PARTICIPANT FLOW:
Groups:
- Straight CPAP: Patients randomized to straight CPAP will receive 10 cm of air pressure, or as determined by the results of polysomnography, for 6 weeks. Following the 6-week visit, patients will be placed on straight CPAP with equipment approved by insurance for an additional 6 weeks.
  Straight CPAP
- Sham CPAP: Patients randomized to sham CPAP will receive 1-2 cm of air pressure for 6 weeks. Following the 6-week visit, patients will be placed on straight CPAP with equipment approved by insurance for an additional 6 weeks.
  Sham CPAP
Period: Overall Study
Arm/Group | Straight CPAP | Sham CPAP
Started | 12 | 10
Completed | 9 | 9
Not Completed | 3 | 1
Not completed — Failure to tolerate CPAP/Sham CPAP | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Straight CPAP | Sham CPAP | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (10.9) | 62.7 (6.3) | 57.2 (10.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity and Race information not collected
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity and race information not collected.
Region of Enrollment [Number; unit: participants] — Population: Region of Enrollment information not collected

OUTCOME MEASURES:

1. Primary Outcome: Change in Leicester Cough Questionnaire Score
Description: Subjects will complete the Leicester Cough Questionnaire at the baseline and 6-week visits. The Leicester Cough Questionnaire comprises 19 items, which assess symptoms, or the impact of symptoms, over the last 2 weeks on a seven-point Likert scale. Scores in three domains (physical, psychological and social) are calculated as a mean for each domain (range 1 to 7). A total score (range 3 to 21) is also calculated by adding the domain scores together. Higher scores indicate better quality of life. The change in Leicester Cough Questionnaire score will be compared between the Straight CPAP and Sham CPAP groups
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Straight CPAP | Sham CPAP
Number analyzed (Participants) | 9 | 9
score on a scale | 6.61 (1.36) | 2.07 (0.98)

2. Secondary Outcome: Change in Cough Frequency
Description: Subjects will wear a Leicester cough monitor for 24 hours at the baseline and 6-week visits, which will record cough frequency during that period. The change in cough frequency from baseline to 6 weeks will be compared between the Straight CPAP and SHAM CPAP groups
Time Frame: Baseline and 6 weeks
Population: Cough monitoring for 24 h at baseline, 6 weeks, and 12 weeks. Due to inadequate duration of cough monitoring data in study patients at baseline (24 hour), comparisons of cough frequency at 6 weeks and 12 weeks between these two groups could not be done in this study.
Arm/Group | Straight CPAP | Sham CPAP
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: 8 Isoprostane Level in Exhaled Breath Condensate
Description: Samples of breath condensate will be collected from study subjects at the baseline and 6-week visits. The 8 isoprostane level from baseline to 6-weeks will be compared between the Straight CPAP and Sham CPAP groups
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Straight CPAP | Sham CPAP
Number analyzed (Participants) | 9 | 9
pg/mL
  Baseline | 4.92 (2.23) | 3.99 (1.89)
  6 weeks | 7.35 (3.47) | 5.04 (2.13)

4. Secondary Outcome: Interleukin-8 (IL-8) Level in Exhaled Breath Condensate
Description: Samples of breath condensate will be collected from study subjects at the baseline and 6-week visits. IL-6 level from baseline to 6-weeks will be compared between the Straight CPAP and Sham CPAP groups
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Straight CPAP | Sham CPAP
Number analyzed (Participants) | 9 | 9
pg/mL
  Baseline | 1.52 (1.41) | 1.02 (0.24)
  6 weeks | 1.00 (0.21) | 1.04 (0.18)

5. Secondary Outcome: Nitrite/Nitrate (NOX) Level in Exhaled Breath Condensate
Description: Samples of breath condensate will be collected from study subjects at the baseline and 6-week visits. NOX level from baseline to 6-weeks will be compared between the Straight CPAP and Sham CPAP groups.
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | Straight CPAP | Sham CPAP
Number analyzed (Participants) | 9 | 9
μmol/L
  Baseline | 3.34 (2.07) | 3.35 (2.81)
  6 weeks | 2.91 (2.32) | 5.26 (0.18)

6. Secondary Outcome: Hydrogen Peroxide (H2O2) Level in Exhaled Breath Condensate
Description: Samples of breath condensate will be collected from study subjects at the baseline and 6-week visits. H2O2 level from baseline to 6-weeks will be compared between the Straight CPAP and Sham CPAP groups
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Straight CPAP | Sham CPAP
Number analyzed (Participants) | 9 | 9
nmol/L
  Baseline | 2458.02 (324.88) | 1714.42 (337.1)
  6 weeks | 1654.07 (239.71) | 1468.04 (143.58)

7. Secondary Outcome: Change in Leukotriene B4 (LTB4) Level in Exhaled Breath Condensate
Description: Samples of breath condensate will be collected from study subjects at the baseline and 6-week visits. The change in LTB4 level from baseline to 6-weeks will be compared between the Straight CPAP and Sham CPAP groups
Time Frame: Baseline and 6 weeks
Population: Due to instability of LTB4 condensate samples stored greater than 3 weeks, LTB4 measurements were not analyzed.
Arm/Group | Straight CPAP | Sham CPAP
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in Gastroesophageal Reflux Disease Quality of Life (GERD-QoL) Questionnaire Score
Description: Subjects will complete the GERD-QoL questionnaire at the baseline and 6-week visits. The GERD-QoL comprises 15 items on a five-point Likert scale; lowest possible score (0) = no symptoms, greatest possible score (75) = worst symptoms. The change in GERD-QoL score will be compared between the Straight CPAP and Sham CPAP groups
Time Frame: Baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Straight CPAP | Sham CPAP
Number analyzed (Participants) | 9 | 9
score on a scale | 9.4 (22.25) | 6.3 (6.7)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Straight CPAP | Sham CPAP
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9
Other Adverse Events (participants affected / at risk) | 0/9 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-01): https://cdn.clinicaltrials.gov/large-docs/30/NCT03172130/Prot_SAP_000.pdf